CLINICAL TRIAL: NCT04528966
Title: Short and Long-Term Effects of Whole Body Vibration on Spasticity and Motor Performance in Children With Hemiparetic Cerebral Palsy
Brief Title: Effects of WBV in Children With Hemiparetic CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fatih Tekin, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PamukkaleUni
Record Dates: First submitted 2020-02-15; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Cerebral Palsy; Whole Body Vibration; Spastic Hemiplegia; Motor Performance
Keywords: Cerebral Palsy; Spasticity; Motor Performance; Whole-Body Vibration; Conventional Physical Therapy
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Group that have received whole-body vibration treatment in addition to conventional physiotherapy
  Interventions: Other: Whole-Body Vibration; Other: Conventional Physiotherapy
- Control group (Active Comparator): Group that have received conventional physiotherapy only
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Whole-Body Vibration — Whole-Body Vibration Treatment for 3 sessions in a week for 8 weeks. Each sessions takes 15 minutes.
  Arms: Treatment Group
Other: Conventional Physiotherapy — conventional physiotherapy for 2 sessions in a week for 8 weeks. Each sessions takes 45 minutes.

SUMMARY:
The aim of this study was to investigate short and long-term effects of Whole Body Vibration therapy on spasticity and motor performance in children with hemiparetic cerebral palsy in addition to conventional physiotherapy.

Twenty-six patients undergoing conventional physiotherapy in a private rehabilitation center were included in the study. Patients were randomized to treatment and control groups. Study was completed with a total of 22 cases (11 for each group). At the beginning of the study, cases were evaluated with Gross Motor Function Measure-88, LEGSys Spatio-Temporal Gait Analyzer, SportKAT550tm Portable Computerized Kinesthetic Balance Device and Modified Ashworth Scale. Cases in the treatment group were treated with Compex-Winplate for 8 weeks, 3 times a week, 15 minutes a day in one session. All cases were reevaluated immediately after the treatment and 12 weeks after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with hemiparetic CP
* patients were followed-up and treated by a special rehabilitation center
* aged between 6-18 years
* patients could walk independently without using assistive devices

Exclusion Criteria:

* any other neurological diseases
* cooperation problems
* visual or auditory disability

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Gross Motor Functions assessed by Gross Motor Function Measure-88 | 1 year
  Gross Motor Function Measure-88 (GMFM-88) will be used to determine the functional skill level. GMFM-88 For a child with Cerebral Palsy (CP) with 5 sub-dimensions, lying, rolling (Dimension A), sitting (Dimension B), kneeling trunk control (Dimension C), standing (Dimension D) and walking activities (Dimension E) ) and measures the rate of realization of activities. Accordingly, the multiplication of the score obtained by the patient in each dimension by the division of the maximum score that can be obtained in that dimension by 100 indicates the percentage score obtained for that dimension. The total GMFM-88 score is obtained by dividing the sum of the scores obtained from the dimensions by 5 (Dimension A-E). As the score obtained increases, the level of performing gross motor skills of the patient with CP also increases.
Gait Parameters Assessed Using Modified Timed Up and Go Test by LegSys Spatio-Temporal Gait Analysis System | 1 year
  The gait performance of the cases was evaluated with the spatio-temporal gait analyzer called LEGSys developed by BioSensics. The device consists of two sensors. The sensors are placed between the ankle joint and the knee joint of the patient to be tested, with the aid of velcro, closer to the ankle. The device is controlled from the computer with its own software and sends the raw data it collects to the computer instantly via Bluetooth. The software analyzes the raw data it receives from the device and converts it into results.
  For the evaluation, the Modified Timed Up and Go Test (MTUG), which was also supported by the device, was used. MTUG is a tool that assesses one's mobility and requires both static and dynamic balance. This test is a scale of the World Health Organization model of International Classification of Functioning Disability and Health. The test was repeated 2 times and the mean time was recorded.
Balance Skills Assessed by SportKAT 550 | 1 year
  The balance skills of the subjects were evaluated with SportKAT 550 portable computerized kinesthetic balance device, which was developed to evaluate the static and dynamic balance, which gives sensitive information about postural stability. The data obtained from the device are quantitative and objective.
  The Balancing Index measures a person's ability to hold the platform near the reference position. The scores ranges from 0 to 6000. Low score indicates good performance. For static tests, a PSI level of 5, a score of 250 or less, is excellent. A score of 500 is good. A score of over 750 indicates a defect in the equilibrium system and indicates a risk of falling. However, excellent, good or at-risk values vary from individual to individual.
Spasticity Assessed by Modified Ashworth Scale | 1 year
  It is a widely used scale for the evaluation of spasticity. If the muscle to be tested is a flexor muscle, the joint is maximally extended in about one second while in the maximum flexion position. If the muscle to be tested is an extensor muscle, it is started when the joint is at maximum extension and maximized in one second. Scoring from 0 to 4 (0, 1, 1+, 2, 3, 4) is made according to resistance taken from muscle. It is also seen that various studies have scored "0,1,2,3,4,5" for MAS. The validity and reliability of this scoring method in hemiparetic individuals has been showed with different studies. 0 means no increase in muscle tone and 5 means that the limb is in a rigid position.
  In this study, knee extensors and ankle plantar flexors' spasticities were evaluated and total spasticity score was calculated by summing up one by one. Similarly, upper extremity total spasticity score was calculated by evaluating elbow flexors, forearm pronators and wrist flexors.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Tekin, PT PhD, Principal Investigator — Research Assistant
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No